CLINICAL TRIAL: NCT02262026
Title: A Phase One Study Investigating the Tolerability and Effects of AZD0530 on Functional Neuroimaging Responses in Individuals With or Without a Family History of Alcoholism
Brief Title: The Tolerability and Effects of AZD0530 in Individuals With or Without a Family History of Alcoholism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1503015528
Record Dates: First submitted 2014-10-01; First posted 2014-10-10 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — saracatinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- FHP; 125mg AZD0530, then 50mg AZD0530, then placebo (Experimental): Family History positive for alcoholism will take place in blinded testing of 125 mg, then 50 mg, then placebo separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHP; 125mg AZD0530, then placebo, then 50mg AZD0530 (Experimental): Family History positive for alcoholism will take place in blinded testing of 125 mg, then placebo, then 50mg separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHP; 50mg AZD0530, then 125mg AZD0530, then placebo (Experimental): Family History positive for alcoholism will take place in blinded testing of 50mg, then 125mg, then placebo separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHP; 50mg AZD0530, then placebo, then 125mg AZD0530 (Experimental): Family History positive for alcoholism will take place in blinded testing of 50mg, then placebo, then 125mg separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHP; placebo, then 50mg AZD0530, then 125mg AZD0530 (Experimental): Family History positive for alcoholism will take place in blinded testing of placebo, then 50 mg, then 125 mg separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHP; placebo, then 125mg AZD0530,then 50mg AZD0530 (Experimental): Family History positive for alcoholism will take place in blinded testing of placebo, then 125 mg, then 50 mg separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHN; 125mg AZD0530, then 50mg AZD0530, then placebo (Active Comparator): Family History negative for alcoholism will take place in blinded testing of 125 mg, then 50 mg, then placebo separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHN; 125mg AZD0530, then placebo, then 50mg AZD0530 (Active Comparator): Family History negative for alcoholism will take place in blinded testing of 125 mg, then placebo, then 50mg separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHN; 50mg AZD0530, then 125mg AZD0530, then placebo (Active Comparator): Family History negative for alcoholism will take place in blinded testing of 50mg, then 125mg, then placebo separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHN; 50mg AZD0530, then placebo, then 125mg AZD0530 (Active Comparator): Family History negative for alcoholism will take place in blinded testing of 50mg, then placebo, then 125mg separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHN; placebo, then 50mg AZD0530, then 125mg AZD0530 (Active Comparator): Family History negative for alcoholism will take place in blinded testing of placebo, then 50 mg, then 125 mg separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo
- FHN; placebo, then 125mg AZD0530, then 50mg AZD0530 (Active Comparator): Family History negative for alcoholism will take place in blinded testing of placebo, then 125 mg, then 50 mg separated by 1 week for each test
  Interventions: Drug: 125 mg AZD0530; Drug: 50 mg AZD0530; Drug: Placebo

INTERVENTIONS:
Drug: 125 mg AZD0530 — Randomized to receive 125 mg of AZD0530
  Other Names: saracatinib; AZD0530
Drug: 50 mg AZD0530 — Randomized to receive 50 mg of AZD0530
  Other Names: saracatinib; AZD0530
Drug: Placebo — Placebo

SUMMARY:
Functional neuroimaging of alcoholism vulnerability: glutamate, reward, impulsivity, and Pavlovian-to-instrumental transfer (PIT), part II Saracatinib

DETAILED DESCRIPTION:
To assess the effect of oral AZ D0530 at various doses on neuroimaging parameters associated with various forms of impulsivity mediated through glutamate-dopamine interactions, as ascertained through functional magnetic resonance imaging. -- --NOTE-- AZD0530 dosage of 50mg was discontinued by manufacturer. Adjustments were made to account for the removal of the 50mg dosage in all arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* Clear History of a father having a history of alcoholism, OR a mother AND another 1st or 2nd degree relative having a history of alcoholism, OR no 1st or 2nd degree relatives with alcoholism or substance abuse

Exclusion Criteria:

1. Current diagnosis of DSM-IV-TR Axis I disorder, or past diagnosis of any substance use disorder or moderate alcohol use disorder
2. Report of psychotic disorder in a 1º relative
3. Auditory or visual impairment that interferes with test taking
4. History of prenatal exposure to alcohol plus currently meeting criteria for features of fetal alcohol syndrome
5. Not speaking English fluently or being a non-native English speaker, or being educated in a primary language other than English >grade 1
6. Mental retardation (Full Scale IQ<70) using 2 WASI subtests for IQ estimate
7. Traumatic brain injury with loss of consciousness > 30 minutes, or concussion in last 30 days
8. Presence or history of any medical/neurologic illness that may affect brain physiology (e.g., epilepsy, Multiple Sclerosis), including focal brain lesion seen on structural MRI (all structural scans are read by a licensed radiologist)
9. Current pregnancy (all females will be tested with urine screens on the day of MRI and prior to each phase of drug treatment)
10. Positive urine screen for the presence of marijuana, cocaine, opiates or breath screen to detect the presence of alcohol, administered at each lab visit.
11. Inability to comprehend the consent form appropriately
12. Ferromagnetic metal devices, clips or fragments in body (orbital x-ray performed if needed).
13. Current use (within 30 days of screening) of specific psychoactive medications (e.g., typical neuroleptics, narcotic analgesics, antiparkinsonian medications, systemic corticosteroids, or medications with significant central anticholinergic activity, etc.). Current use of warfarin.
14. Current use of the following medications (CYP3A4 substrates whose metabolism may be slowed by AZD0530): carbamazepine, colchicine, cyclosporine, disopyramide, fluticasone, quinidine, vinblastine, vincristine, nifedipine. Patients taking sildenafil, tadalafil, and vardenafil will be advised to stop taking these medications for the duration of the trial. Patients cannot take the following drugs which inhibit the CYP3A4 isoenzyme: cimetidine, cyclosporine, danazol, fluconazole, grapefruit juice, HIV protease inhibitors, itraconazole, ketoconazole, macrolides, miconazole, nefazodone, omeprazole, ritonavir, and verapamil, aromatase inhibitors, docetaxel
15. Neutropenia defined as absolute neutrophils count of <1,500/microliter.
16. Thrombocytopenia defined as platelet count <100x103/microliter.
17. AST, ALT, total bilirubin >1.5 times upper normal; serum creatinine, >2 time upper normal limit, total bilirubin>1.5 times ULN; Serum creatinine >2.0 times ULN.
18. History of interstitial lung disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
BOLD activation during A1 phase | 4 Hours post medication administration
  BOLD activation during the A1 phase of the MRI Monetary Incentive Delay task

SECONDARY OUTCOMES:
BOLD signal activation in the anterior cingulate cortex(ACC) | 4 Hours post medication administration
  BOLD signal activation in the anterior cingulate cortex (ACC) observed during False Alarms of the GoNoGo Task

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey D Pearlson, MD, Principal Investigator — Yale University
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02262026/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02262026/ICF_001.pdf